CLINICAL TRIAL: NCT03970707
Title: Investigation on Recovery Kinetics After the Use of Small Sided Games With a Small and Large Number of Players and Large Pitch Area
Brief Title: Recovery Kinetics After the Use of Small Sided Games With a Small and Large Number of Players and Large Pitch Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: REKI-SSG
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Sided Games in Soccer Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Small Number of Players training protocol A (Experimental): Small Sided Game: 4 vs 4
  Interventions: Other: Small Number of Players training protocol A
- Large Number of Players training protocol B (Experimental): Small Sided Game: 8 vs 8
  Interventions: Other: Large Number of Players training protocol B
- Control (No Intervention): No training protocol will be performed, the participants will perform only the measurements for performance and muscle damage and neuromuscular fatigue

INTERVENTIONS:
Other: Small Number of Players training protocol A — 8 participants each side game (4vs4), size of pitch area 25*20 m. In total, 6 consecutive 4-minutes bouts interspersed by a 3-minutes rest between each bout will be executed.
  Arms: Small Number of Players training protocol A
Other: Large Number of Players training protocol B — 16 participants each side game (8vs8), size of pitch area 25*20 m. In total, 3 consecutive 8-minutes bouts interspersed by a 1-minutes rest between each bout will be executed.
  Arms: Large Number of Players training protocol B

SUMMARY:
Soccer is an intermittent sport in which the aerobic and anaerobic capacity of the players are both essential. Elite football players perform an average of 150-250 short and intense movements during a match, demonstrating the significant contribution of the anaerobic energy system. Sided-games is a tool to enhance the performance of the aerobic and anaerobic system. This training includes actions such as sprinting, changes of direction, accelerations, decelerations, jumps, and shooting, characterized by a strong eccentric component. Eccentric actions are associated with exercise-induced muscle damage (EIMD). Nevertheless, to date, EIMD responses following a session of sided games training have not yet been investigated. Therefore, the present study aims to examine the speed of recovery after training with a large-dimension pitch area with a small and large number of athletes in football.

DETAILED DESCRIPTION:
Football is an intermittent sport that includes actions of variable intensities and combines elements of physical fitness with technical and tactical skills. The game is characterized by a combination of several short-term movements such as jumps and change of direction. Typically, a player in a soccer game changes his kinetic situation every 4-6 seconds. The mean and maximum heart rate during the fight is approximately 85% and 98% of the maximum heart rate, respectively, while the average oxygen uptake is 70% of the maximum, proving that the aerobic system contributes significantly during the game. In addition, the lactic acid value in the blood ranges from 2 to 14 mM, which proves that also the anaerobic energy system contributes significantly during a game. Based on the above, the training of soccer players must meet the physiological and physiological requirements of the game.

There are two approaches to developing fitness. In the first, there is a distinction between fitness training technical skills and tactics, while the second attempts to achieve all of them at the same time, and for that purpose, the sided games are used. The first approach refers to the literature as a traditional form of physical fitness training and contains the ball and run exercises. It is part of the training unit and separates the physical conditioning from the technique and tactics, resulting in longer training time. Moreover, although this training achieves the necessary physiological adaptations, the piece of game specialization is missing. For this reason, coaches have been interested in the sided games with restrictions, combining physical, technical, and tactical elements. The coach can modify these games to achieve the training goal each time. During training with racing blocks, a similar or even higher heart rate has been observed on soccer players compared with the short-term intermittent exercise. The intensity of the exercise on the sided games is controlled by several variables that the coach can modify according to the training goal. Many variables can affect the training load such as pitch area, the number of players, and other restrictions (e.g., goalkeepers, contact limitation, etc.). In the application of sided games with large dimension and a small number of players, the maximum heart rate can reach 84-90% while with a large number of players it can reach 84-88%. There is a lack of references regarding rehabilitation after the implementation of sided games, and especially after the execution of large-dimension pitch area with a small and large number of athletes. The aim of the proposed study is, therefore, to examine the speed of recovery after training with a large-dimension pitch area with a small and large number of athletes in football.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of any musculoskeletal injury for at least 6 months prior to the study
2. No use of any drugs or ergogenic supplements for at least 6 months prior to the study
3. Absence of regular soccer training for the last 3 years

Exclusion Criteria:

1. Any recent incidence of musculoskeletal injury
2. Use of any drugs or ergogenic supplements for the last 6 months
3. Regular soccer training for the last 3 years-

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences in changes in creatine kinase (CK) between the two training protocols | Pre-protocol, Day 1, Day 2, Day 3
  Creatine kinase (CK) is a muscle damage marker
Differences in changes in delayed onset of muscle soreness (DOMS) between the two training protocols | Pre-protocol, Day 1, Day 2, Day 3
  Delayed onset of muscle soreness (DOMS) is a muscle damage marker
Differences in changes in maximal concentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal concentric strength is used as a muscle damage marker
Differences in changes in maximal eccentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal eccentric strength is used as a muscle damage marker

SECONDARY OUTCOMES:
Differences in changes in countermovement jump between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Countermovement jump is used as a performance marker
Differences in changes in Repeated Sprint Ability (RSA) between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Repeated Sprint Ability (RSA) is a performance marker
Differences in changes in maximal concentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal concentric strength is used as a performance marker
Differences in changes in maximal eccentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal eccentric strength is used as a performance marker
Differences in changes in maximal isometric strength between the two training protocols | Baseline, Hour 1, Hour 2, Hour 3
  Maximal isometric strength is used as a neuromuscular fatigue marker

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, PhD, Principal Investigator — DPESS, School of Physical Education, Sport & Dietetics, University of Thessaly
Locations (1):
- SmArT LABORATORY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES, UNIVERSITY OF THESSALY, Trikala, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohr M, Krustrup P, Bangsbo J. Match performance of high-standard soccer players with special reference to development of fatigue. J Sports Sci. 2003 Jul;21(7):519-28. doi: 10.1080/0264041031000071182. PMID 12848386
- [Background] Ade JD, Harley JA, Bradley PS. Physiological response, time-motion characteristics, and reproducibility of various speed-endurance drills in elite youth soccer players: small-sided games versus generic running. Int J Sports Physiol Perform. 2014 May;9(3):471-9. doi: 10.1123/ijspp.2013-0390. Epub 2014 Feb 7. PMID 24509482
- [Background] Fatouros IG, Chatzinikolaou A, Douroudos II, Nikolaidis MG, Kyparos A, Margonis K, Michailidis Y, Vantarakis A, Taxildaris K, Katrabasas I, Mandalidis D, Kouretas D, Jamurtas AZ. Time-course of changes in oxidative stress and antioxidant status responses following a soccer game. J Strength Cond Res. 2010 Dec;24(12):3278-86. doi: 10.1519/JSC.0b013e3181b60444. PMID 19996787
- [Background] Hill-Haas SV, Dawson B, Impellizzeri FM, Coutts AJ. Physiology of small-sided games training in football: a systematic review. Sports Med. 2011 Mar 1;41(3):199-220. doi: 10.2165/11539740-000000000-00000. PMID 21395363
- [Background] Owen AL, Wong DP, Paul D, Dellal A. Physical and technical comparisons between various-sided games within professional soccer. Int J Sports Med. 2014 Apr;35(4):286-92. doi: 10.1055/s-0033-1351333. Epub 2013 Sep 10. PMID 24022576